CLINICAL TRIAL: NCT03684746
Title: Innovation Adoption in Medical Robotic Surgery: Case of Royal Bournemouth Hospital
Status: Completed | Type: Observational
Sponsor: Bournemouth University (Other)
Collaborators: Royal Bournemouth Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1718/IRASMSE/1
Record Dates: First submitted 2018-06-29; First posted 2018-09-26 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Staff Attitude

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medial Experts: Including doctors- surgeons - consultants
  Interventions: Other: No Intervention
- Care specialist: including nurses - before/after care staff
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — It is an observational Study with staff

SUMMARY:
This research sets to address two key areas. The first is identified by the researcher in academic literature that there is a lack of a comprehensive innovation adoption model in UK National Health System (NHS), specifically for Medical Robotic Surgery. Existing frameworks are mainly developed in the US or in other fields. The second problem was identified by surgeons involved in Robotic Surgery in Royal Bournemouth Hospital (RBH). The project started by offering RBH a deeper understanding of the innovation adoption process, issues and development of an adapted innovation model, however after our initial meeting with the Surgical Director and his team, it was clear that one the main areas RBH was keen for us to investigate, was the communication pathway of all stakeholders involved in robotic surgery adoption. They were concerned that key staff dealing with patients undergoing medical robotic surgery were uninformed about the technology and process which can impact patients' experience and staff communication.

The research will develop a comprehensive innovation adoption model for robotic surgery (and similar medical innovation) in NHS. Currently there are no models adapted to NHS UK structure and requirements. This model will assist the NHS to understand and evaluate any innovation adoption process within the NHS and to avoid future innovation adoption failure.

The case example will Identify the communication pathway and key stakeholders in RBH for the process of Gastrointestinal Robotic Surgery, evaluation of stakeholders' knowledge and needs and further proposing ways to improve adoption and increase knowledge. NHS can use the proposed communication pathway to identify stakeholders that need to be informed, trained and communicated to, in any innovation adoption process within NHS.

ELIGIBILITY:
Inclusion Criteria:

Being involved with conducting Robotic Surgery or caring for patients undergoing Robotic Surgery

Exclusion Criteria:

-

As this study is recruiting staff, and there is no medical intervention, the eligibility criteria is basic.

Max Age: 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Medical experts and hospital staff involved directly on indirectly in Robotic Surgery at the NHS site - these individuals will have the necessary knowledge to contribute to this study.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Surgical Innovation Framework | 6 months
  To develop a 'Surgical Innovation Framework' through discussion with surgeons, medical experts and staff at the research site. This framework would then be of use to other medical/surgical areas within the NHS, as there is currently no model adapted to the NHS' needs and requirements. The research will increase knowledge and enable better communication.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Bournemouth Hospital, Bournemouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No
I am not planning to share any data with other researchers.